CLINICAL TRIAL: NCT06324435
Title: Apremilast for Alcohol Use Disorder Treatment in Women and Men
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Office of Research on Women's Health (ORWH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2000037439; 1U54AA027989-01 (NIH)
Record Dates: First submitted 2024-03-14; First posted 2024-03-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — apremilast

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Apremilast (Experimental): Apremilast (60mg/day). Administered orally twice daily at 8:00 AM and 8:00 PM while titrating to the full dose. Titration schedule: Day 1 10mg AM; Day 2 10mg AM, 10mg PM; Day 3 10mg AM, 20mg PM; Day 4 20mg AM, 20mg PM; Day 5 20mg AM, 30mg PM; Day 6 30mg AM, 30mg PM. Once at steady state, administration is orally twice daily at 8:00 AM (30mg) and 8:00 PM (30mg).
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — 60mg/day
  Other Names: Otezla

SUMMARY:
For this protocol, the investigators plan to collect pilot data to evaluate apremilast (60mg/day) in adults with Alcohol Use Disorders (AUD).

DETAILED DESCRIPTION:
This study is a Phase 1 open-label design to evaluate apremilast (60mg/day) in adults meeting criteria for DSM-5 alcohol use disorders (n=10).

Eligibility screening consists of an intake session and a physical exam. Subjects meeting eligibility criteria will be assigned to apremilast (60mg/day). Titration to steady state medication levels will occur over 6 days (Day 1-6). Subjects will then complete two laboratory sessions and a cue-reactivity session (Days 7-21). During each laboratory session, personalized imagery (within- subject factor, either stress or neutral/relaxing, order counterbalanced) will precede a 2-hour alcohol self-administration period.

No taper medication is needed. Following the medication discontinuation (Day 22), subjects will be contacted to assess any side effect from discontinuing medication (Day 36).

Adverse events are evaluated at each study appointment and will be tabulated.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 21-65.
4. Able to read and write English
5. Meets DSM-5 criteria for current (past 6 months) AUD
6. Drinking criteria: males - drinks > 14 drinks per week and exceeds 4 drinks per day at least twice per week; females - drinks > 7 drinks per week and exceeds 3 drinks per day at least twice per week. They must meet drinking criteria during a consecutive 30-day period prior to baseline.
7. Laboratory sessions will be scheduled such that subjects will not have major responsibilities on the following day which might limit drinking during the self-administration session (e.g., job interview, exam)
8. Able to take oral medications and willing to adhere to a medication regimen.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Subjects with any significant current medical conditions (neurological, cardiovascular, endocrine, thyroid, renal, liver), seizures, delirium or hallucinations, or other unstable medical conditions, including HIV
2. Current DSM-5 substance use disorder (other than AUD or tobacco use disorder)
3. A positive test result at intake appointment on urine drug screens conducted for illicit drugs.
4. Past 30-day use of psychoactive drugs may be included at the discretion of the study MD as long as the concurrent treatment does not compromise the study integrity by virtue of its type, duration, or intensity.
5. Women who are pregnant or nursing, or fail to use one of the following methods of birth control unless she or her partner is surgically sterile or she is postmenopausal (hormone contraceptives [oral, implant, injection, patch, or ring], contraceptive sponge, double barrier [diaphragm or condom plus spermicide], or IUD)
6. Suicidal, homicidal, or evidence of current (past 6 months) mental illness such as schizophrenia, bipolar disorder or major depression, or anxiety disorders
7. Only one member per household can participate in the study
8. Specific exclusions for administration of apremilast not already specified include: known hypersensitivity to apremilast; cytochrome P450 enzyme inducers (e.g., rifampin, phenobarbital, carbamazepine, phenytoin).
9. Drugs that may influence study outcomes (e.g., disulfiram, naltrexone, acamprosate, anticonvulsants).
10. Subjects likely to exhibit clinically significant alcohol withdrawal during the study. We will exclude subjects who a) have a history of perceptual distortions, seizures, delirium, or hallucinations upon withdrawal, or b) have a score of > 8 on the Clinical Institute Withdrawal Assessment scale at intake appointments.
11. Subjects who have taken any investigational drug within 4 weeks immediately preceding admission to the treatment period.
12. Participation within the past 8 weeks in other studies that involve additive blood sampling and/or interventional measures that would be considered excessive in combination with the current application.
13. Those currently in treatment for alcohol use, individuals with a history of serious withdrawal, and individuals who have repeatedly undergone alcohol detoxification.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol Consumption | 120 minutes
  Means mls of alcohol consumed during 120 minute alcohol self-administration sessions with personalized stress imagery vs neutral/relaxing imagery taking place at steady state.

CONTACTS AND LOCATIONS:
Overall Officials: Sherry McKee, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No